CLINICAL TRIAL: NCT03460821
Title: Validation of a German Translation and Cultural Adaptation of the Addenbrooke's Cognitive Examination III
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and operative Intensive Care Medicine (CCM, CVK), Charite University, Berlin, Germany
Other Study IDs: ACE-III
Record Dates: First submitted 2018-02-27; First posted 2018-03-09 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Neurocognitive Dysfunction
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Employees: Male and female employees (≥ 18 years of age) of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité Universitätsmedizin Berlin experienced in the field of neurocognitive testing: residents, specialist physician for anesthesiology, senior physicians, medical students engaged in research projects

SUMMARY:
The aim of the entire project was to perform a translation and cultural adaptation of the Addenbrooke's Cognitive Examination - III (ACE-III), adhering to the Translation and Cultural Adaptation of Patient Reported Outcomes Measures-Principles of Good Practice, in order to make it available to German clinicians.

Part of the translation process is the cognitive debriefing which will be performed as a survey which rates the applicability of every single item as well as of the entire Addenbrooke's Cognitive Examination - III tool.

DETAILED DESCRIPTION:
The recent demographic developments have drastically increased the importance of developing applicable approaches to the diagnostics of dementia and the general evaluation of cognitive function. Many different tests were developed to thoroughly evaluate neurocognitive function.

The Addenbrooke's Cognitive Examination, developed in 2000, was one such tests and has served as an open source neurocognitive examination tool ever since. The current version is the Addenbrooke's Cognitive Examination III (ACE-III). The aim was to develop a tool that would be able to identify dementia in its early stages and also to differentiate between the different types of dementia.

In order to achieve reliable results, cognitive tests should be conducted in a familiar language and draw from the cultural background a participant is familiar with. The ACE-III and all its predecessors were developed in English and for an English-speaking cultural background, not directly applicable to the typical German patient. This made it necessary to perform not only a verbatim translation of test contents, but also to appropriately adapt the test content to reflect the cultural background of the typical German patient. The International Society For Pharmacoeconomics and Outcomes Research (ISPOR) - Task Force for Translation and Cultural Adaptation has developed the "Translation and Cultural Adaptation of Patient Reported Outcomes Measures-Principles of Good Practice", to ensure a consistent and rigorous methodology in the process of translating and adapting patient-reported outcomes measures.

The Principles of Good Practice consist of ten steps:

1. Preparation
2. Forward Translation
3. Reconciliation
4. Back Translation
5. Back Translation Review
6. Harmonization
7. Cognitive Debriefing
8. Review of Cognitive Debriefing Results and Finalization
9. Proofreading
10. Final Report

ELIGIBILITY:
Inclusion Criteria:

* Male and female employees of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité Universitätsmedizin Berlin (residents, specialist physician for anesthesiology, senior physicians, medical students engaged in research projects)

  .- ≥ 18 years of age
* Experience in the field of neurocognitive testing

Exclusion Criteria:

* Insufficient knowledge of the German language

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female employees (≥ 18 years of age) of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité Universitätsmedizin Berlin experienced in the field of neurocognitive testing
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of respondents who rate the questionnaire as "applicable" or "not applicable" | Up to one month
  The overall applicability of the German translation will be evaluated on a scale from 0 (not applicable) to 5 (applicable without any restrictions). A priori, a score of ≥ 4 was defined as indicating applicability. The overall applicability will be judged by the amount of survey respondents rating the entire battery as applicable, in relation to the total number of respondents.

SECONDARY OUTCOMES:
Percentage of the items which are rated as "applicable" or "not applicable" | Up to one month
  Description: The applicability of each individual item will be evaluated on a scale from 0 (not applicable) to 5 (applicable without any restrictions). A priori, a score of ≥ 4 was defined as indicating applicability. The overall applicability will be judged by the amount of survey respondents rating the entire battery as applicable, in relation to the total number of respondents
Mean/Median applicability of the entire survey | Up to one month
  Mean/Median applicability of the entire survey will be calculated using the applicability ratings of the entire survey (as described above)
Frequency of limiting factors of the entire Addenbrooke's Cognitive Examination - III questionnaire | Up to one month
  If participants rate the entire survey as not applicable (rating < 4) they are asked to choose a limiting factor from a predefined list. The frequency with which every limiting factor is mentioned is compiled to evaluate its impact on the entire survey
Frequency of limiting factors of the single items | Up to one month
  If participants rate an item as not applicable (rating < 4) they are asked to choose a limiting factor from a predefined list. The frequency with which every limiting factor is mentioned is compiled to evaluate its impact on the entire survey.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operaitve Intensive Care Medicine, Campus Charite Mitte (CCM) and Campus Virchow - Klinikum, Charite - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No